CLINICAL TRIAL: NCT04218916
Title: The Efficacy and Safety of Rhodiola Rosea in Patients With Coronary Microvascular Disease
Brief Title: Rhodiola Rosea for Coronary Microvascular Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, MD, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Qilu Hospital
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Coronary Microvascular Disease
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhodiola Rosea Capsule (Experimental)
  Interventions: Drug: Rhodiola Rosea Capsules
- Placebo Capsule (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rhodiola Rosea Capsules — 0.28g per capsule, 0.56g once (2 capsules), three times a day
  Arms: Rhodiola Rosea Capsule
Drug: Placebo — 2 placebo capsules once, three times a day
  Arms: Placebo Capsule

SUMMARY:
To investigate the effects of rhodiola rosea on coronary flow reserve and symptoms in patients with microvascular angina pectoris, and to evaluate adverse drug reactions. Long-term clinical follow-up of 1 to 3 years was conducted to evaluate the effect of rhodiola rosea on long-term adverse cardiovascular events in patients with coronary microvascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Repeated chest pain attacks with typical exertional angina pectoris or resting angina pectoris attacks;
2. Coronary normal or stenosis < 20%;
3. Ischemic depression in ST segment during resting or exercise;
4. Blood flow reserve (CFR) of the anterior descending coronary artery < 2.0;
5. Subjects or their guardians agreed to participate in this study.

Exclusion Criteria:

1. Previous myocardial infarction or PCI or CABG treatment;
2. A history of heart failure or LVEF < 50%;
3. Severe arrhythmia;
4. Myocarditis, Pericardium Disease, Valvular Disease, or Cardiomyopathy;
5. A history of stroke within half a year;
6. Diabetes difficult to control;
7. Refractory hypertension or hypertension accompanied by left ventricular wall thickness > 12 mm;
8. Familial hypercholesterolemia;
9. Takayasu arteritis, Kawasaki disease or coronary artery malformation;
10. Pregnant or nursing, or having the intention to give birth within one year;
11. Hepatic or renal dysfunction;
12. Other diseases which may cause serious risks to patients;
13. Requiring warfarin anticoagulant therapy; Taking potassium channel opener, CCB, ACEI drugs or traditional Chinese medicines;
14. Allergic to contrast agents or blood products;
15. Patients who participated in clinical research of other drugs within 3 months before being selected.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Coronary Flow Reserve | 1 year